CLINICAL TRIAL: NCT05611281
Title: Phase I Randomized, Double-blind, Placebo-controlled, Single Multiple Dosing, Dose Escalation, and Food Effect Study of GS3-007A Oral Liquid in Chinese Healthy Adults
Brief Title: GS3-007a Oral Solution in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: GenSci073-101
Record Dates: First submitted 2022-09-29; First posted 2022-11-10 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2022-10

CONDITIONS: Healthy Subject

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GS3-007 oral liquid (Experimental): 78 subjects: Part 1 SAD 36 subjects: A total of 6 dose groups of 0.4 mg/kg, 0.8 mg/kg, 1.6 mg/kg, 3.2 mg/kg, 4.8 mg/kg and 6.4 mg/kg are planned. Once a day, a total of one dose.
  Part 2 MAD 30 subjects: Three dose groups of 0.8 mg/kg, 1.6 mg/kg and 3.2 mg/kg were planned，The drug was administered once a day for 7 days Part 3 Food effects 12 subjects: Planned in 1.6mg/kg dose group。Once a day, a total of one dose.
  Interventions: Drug: GS3-007 oral liquid or Placebo GS3-007 oral liquid oral medication
- Placebo GS3-007 oral liquid (Placebo Comparator): Part 1 SAD: A total of 6 dose groups of 0.4 mg/kg, 0.8 mg/kg, 1.6 mg/kg, 3.2 mg/kg, 4.8 mg/kg and 6.4 mg/kg are planned. Once a day, a total of one dose.
  Part 2 MAD: Three dose groups of 0.8 mg/kg, 1.6 mg/kg and 3.2 mg/kg were planned，The drug was administered once a day for 7 days
  Interventions: Drug: GS3-007 oral liquid or Placebo GS3-007 oral liquid oral medication

INTERVENTIONS:
Drug: GS3-007 oral liquid or Placebo GS3-007 oral liquid oral medication — The dosage was calculated according to body weight and dose group once a day according to the assigned group.

SUMMARY:
To evaluate the safety and tolerability of GS3-007A in single, multiple, and single oral administration after high-fat meals in Chinese healthy adults.

DETAILED DESCRIPTION:
This is a first-in-human, The major aims of the study are to define the safety profile of this new drug, and to determine a recommended

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects aged 18-45 years (including boundary values), male and female;
* Body mass index: 19-26 kg/m2 (including boundary value), male weight ≥50 kg, female weight ≥45 kg;

Exclusion Criteria:

* Patients with a history of substance abuse and substance dependence;
* Family history of sudden death;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
TEAEs | Part 1:Changes in safety data from baseline 3 days after dosing; Part 2:Changes in safety data from baseline 10 days after dosing; Part 3:Changes in safety data from baseline 6 days after dosing;
  Adverse events during treatment：Number of participants with treatment-related adverse events as assessed by Guidelines for NIA adverse Events and Serious Adverse Events , To evaluate the safety and tolerability of GS3-007A in single, multiple, and single oral administration after high-fat meals in Chinese healthy adults.

SECONDARY OUTCOMES:
PK characteristics | Part 1: Values measured at baseline and within 3 days after dosing; Part 2: Values measured at baseline and within 10days after dosing; Part 3: Values measured at baseline and within 6 days after dosing;
  To evaluate the pharmacokinetic (Peak Plasma Concentration (Cmax)) characteristics of GS3-007A in Chinese healthy adults after single, multiple, and single oral administration of high-fat meals.

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu Xinhua Hospital Affiliated to North Sichuan Medical College, Chengdu, Chengdu, China